CLINICAL TRIAL: NCT01269606
Title: A Trial Comparing the Pharmacokinetic Properties of Insulin Aspart With Fast-acting Insulin Human Following Intravenous Infusion or Intramuscular Injection in Japanese Subjects With Type 1 Diabetes Mellitus
Brief Title: Comparing Insulin Aspart With Fast-acting Insulin Human in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANA-3877; U1111-1117-1353 (Other: WHO); JapicCTI-111383 (Other: JAPIC)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence 1 - IM treatment group (Experimental)
  Interventions: Drug: insulin aspart
- Treatment sequence 2 - IM treatment group (Experimental)
  Interventions: Drug: insulin human
- Treatment sequence 1 - IV treatment group (Experimental)
  Interventions: Drug: insulin aspart
- Treatment sequence 2 - IV treatment group (Experimental)
  Interventions: Drug: insulin human

INTERVENTIONS:
Drug: insulin aspart — At the first treatment visit, a single dose of insulin aspart at 0.2 U/kg via IM (in the muscle) injection is administered. At the second treatment visit, a single dose of fast-acting insulin human at 0.2 IU/kg via IM (in the muscle) injection is administered. Subjects will resume their usual insulin treatment in the wash-out period of 4-28 days between treatment visits.
  Arms: Treatment sequence 1 - IM treatment group
Drug: insulin human — At the first treatment visit, a single dose of fast-acting insulin human at 0.2 IU/kg via IM (in the muscle) injection is administered.At the second treatment visit, a single dose of insulin aspart at 0.2 U/kg via IM (in the muscle) injection is administered. Subjects will resume their usual insulin treatment in the wash-out period of 4-28 days between treatment periods.
  Arms: Treatment sequence 2 - IM treatment group
Drug: insulin aspart — At the first treatment visit, insulin aspart is intravenously infused for 24 minutes, with rate of 1.25 mU/kg/min at constant phase. At the second treatment visit, fast-acting insulin human is intravenously infused for 24 minutes, with rate of 1.25 mIU/kg/min at constant phase. Subjects will resume their usual insulin treatment in the wash-out period of 4-28 days between treatment visits.
  Arms: Treatment sequence 1 - IV treatment group
Drug: insulin human — At the first treatment visit, fast-acting insulin human is intravenously infused for 24 minutes, with rate of 1.25 mIU/kg/min at constant phase. At the second treatment visit, insulin aspart is intravenously infused for 24 minutes, with rate of 1.25 mU/kg/min at constant phase. Subjects will resume their usual insulin treatment in the wash-out period of 4-28 days between treatment periods.
  Arms: Treatment sequence 2 - IV treatment group

SUMMARY:
This trial is conducted in Japan. The aim of the trial is to compare pharmacokinetics (at which rate the body eliminates the substance from the body) of insulin aspart with fast-acting insulin human following intravenous (IV) infusion or intramuscular (IM) injection in Japanese subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Treated with multiple daily insulin injections for at least 12 months
* Current daily basal insulin requirement above or equal to 0.3 U/kg/day
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 10.0%
* Body Mass Index (BMI) 18.0-28.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start (screening)
* Surgery or trauma with significant blood loss (more than 500 mL) within 3 months prior to trial start (screening)
* Subject who smokes more than 10 cigarettes or the equivalent per day
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clearance at steady state (CLss) for IV treatment group | from 180 min to 240 min
Area under the curve (AUC) for IM treatment group | from 0 to 480 min after intramuscular injection

SECONDARY OUTCOMES:
Area under the curve (AUC) for IM treatment group | from 0 minutes to infinite time after intramuscular injection
Steady state concentration (Css) for IV treatment group | from 180 min to 240 min
Hypoglycaemic episodes | from screening (visit 1) to follow-up visit (2-21 days after last trial product administration)
Adverse Events (AEs) | from first trial related activity to follow-up visit (2-21 days after last trial product administration)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Fukuoka, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com